CLINICAL TRIAL: NCT03860792
Title: Therapeutic Diets in Alzheimer's Disease
Acronym: TDAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Russell Swerdlow, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00143457
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcomes assessors are masked from participant group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (Experimental): Study partners will be instructed to assist participants in adherence to a 1:1 ketogenic diet (approximately 70% fat, <10% carbohydrate, and 20% protein as energy). The diet will encourage ≥4 servings of non-starchy vegetables and 1/2 cup of berries daily. Participants will be provided an emulsified medium chain triglyceride supplement with a target intake of 1-2 tablespoons per day and micronutrient supplements consisting of multivitamin, vitamin D, calcium, and phosphorus. After the 3-month ketogenic diet, participants will complete a 1-month washout period in which they halt adherence to the ketogenic diet and resume their normal diet.
  Interventions: Behavioral: Ketogenic Diet
- Therapeutic Lifestyles Changes Diet (Active Comparator): Study partners will be instructed to assist participants in adherence to the Therapeutic Lifestyles Changes diet. The diet consists of 20-35% fat, 50-60% carbohydrate, and ~15% protein as energy. Fat intake will comprise <7% saturated fat, ≤20% monounsaturated fat, and ≤10% polyunsaturated fat as total energy. Cholesterol consumption will be ≤200mg per day. Participants are encouraged to eat ≥2 servings of fruit and ≥5 servings of vegetables per day.
  Interventions: Behavioral: Therapeutic Lifestyles Changes Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — Three-month 1:1 ketogenic diet intervention (approximately 70% fat, <10% carbohydrate, and 20% protein).
  Arms: Ketogenic Diet
Behavioral: Therapeutic Lifestyles Changes Diet — Three-month diet intervention that is low in fat and cholesterol, high in fruits, vegetables, and whole grains, and moderate in protein.
  Arms: Therapeutic Lifestyles Changes Diet

SUMMARY:
By doing this study, researchers hope to learn how the ketogenic and Therapeutic Lifestyles Changes diets affect cognition in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD by current McKhann et al. criteria
* CDR global score of 0.5 or 1
* Agreed cooperation from an appropriate study partner
* Speaks English as primary language
* Age 50 to 90
* No medication changes within the past 30 days

Exclusion Criteria:

* Resides in a nursing home or dementia special care unit, or cannot control diet
* A potentially confounding serious medical risk including insulin-requiring diabetes, cancer requiring chemotherapy or radiation within the past 5 years, or a recent cardiac event (i.e. heart attack, angioplasty, etc.)
* Participating in another clinical trial or using an investigational drug or therapy within 30 days of the Screening Visit
* A history of renal stones

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance on the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADASCog11) | Baseline, 12 Weeks
  Cognitive performance will be assessed by a psychometrician using the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADASCog11). The ADAS-Cog is an Alzheimer's disease specific, multi-domain cognitive assessment scored from 0-70 points with higher scores indicating poorer cognitive performance.
Change in cognitive performance on the Mini-Mental State Exam (MMSE) | Baseline, 12 Weeks
  Global cognitive performance will be assessed by a psychometrician using the Mini-Mental State Exam (MMSE). The MMSE is a brief cognitive questionnaire with a maximum score of 30 points where higher scores indicate better cognitive performance.
Change in cognitive performance on the Logical Memory Test (LMT) | Baseline, 12 Weeks
  The Logical Memory, subtest of the WMS-R is a standardized assessment of narrative episodic memory. A short story is orally presented, and the examinee is asked to recall the story immediately.
Change in cognitive performance by Stroop test | Baseline, 12 Weeks
  Reaction time and accuracy will be assessed by a psychometrician using the Stroop test.
Change in Clinical Dementia Rating (CDR) | Baseline, 12 Weeks
  The Clinical Dementia Rating is a 5-point scale (CDR 0, 0.5, 1, 2, and 3) used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias. CDR 0 indicates no dementia and higher values indicate more severe dementia. The scores of all six domains are averaged to form a global CDR score. Change in score from baseline to 3 months will be assessed.

SECONDARY OUTCOMES:
Change in cerebral concentration of N-Acetylaspartate (NAA) | Baseline, 12 Weeks
  Concentration of cerebral N-Acetylaspartate is measured using magnetic resonance spectroscopy in a 3T clinical scanner.
Change in blood platelet mitochondrial function | Baseline, 6 Weeks, 12 Weeks
  Cytochrome c oxidase activity of blood platelets will be determined as a pseudo first order-rate constant (sec-1/mg protein) by measuring the oxidation of reduced cytochrome c at 550 nm.
Change in self-reported symptoms by study partner | Baseline, 6 Weeks, 12 Weeks
  Severity of symptoms will be measured via a self-reported symptoms questionnaire, answered by participant study partners.

OTHER OUTCOMES:
Change in blood ketone levels induced by ketogenic diet | Baseline, 6 Weeks, 12 Weeks
  We will measure serum beta-hydroxybutyrate levels.
Proportion of days positive for urinary ketone production | Daily for 90 days (the length of the diet intervention)
  Participants will measure and report daily urinary ketone status using Ketostix (Bayer, Germany).
Dietary intake characterization prior to and after ketogenic diet initiation | Baseline, 6 Weeks, 12 Weeks
  Changes in food and nutrient intake will be assessed by monthly 3-day food records completed by participant study partners.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Science Unit, Fairway, Kansas, United States

IPD SHARING:
Plan to Share IPD: No